CLINICAL TRIAL: NCT02020356
Title: Impact of Music Therapy on Prescription of Neuroleptics in Alzheimer's Disease ou Related Symptoms Associated With Disruptive Behaviours.
Brief Title: Music Therapy in Alzheimer's Disease
Acronym: PRE-MUSICAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/12/0385; AOL 2012 (Other Grant/Funding Number: Local funding)
Record Dates: First submitted 2013-05-30; First posted 2013-12-24 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Alzheimer's Type Dementia
Keywords: Alzheimer's disease; Neuroleptics; Music therapy
MeSH Terms: conditions — Alzheimer Disease | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy (Experimental): "U" sequence: the musical sequence lasts 20 minutes and is made up of several phases that progressively induce a relaxed state in the patient. The phase of maximum relaxation is followed by a stimulating phase.
  Interventions: Behavioral: Music therapy
- Placebo (Placebo Comparator): Interview with an occupational activity (such as discussion of personal pictures or news) with the caregiver in charge of music therapy sessions with the same period.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Music therapy — "U" sequence: the musical sequence lasts 20 minutes and is made up of several phases that progressively induce a relaxed state in the patient. The phase of maximum relaxation is followed by a stimulating phase.
  Arms: Music therapy
Behavioral: Placebo — Interview with an occupational activity (such as discussion of personal pictures or news) with the caregiver in charge of music therapy sessions with the same period.
  Arms: Placebo

SUMMARY:
The primary purpose of the protocol is to demonstrate that the use of music therapy may make it possible to discontinue at least one of neuroleptic treatment in patients with AD or related symptoms complicated by behavioral disorders such as agitation and aggressiveness evaluated using the Neuropsychiatric Inventory (NPI).

The study hypothesis is that music therapy may have a positive impact on patients with AD complicated by behavioral disorders by reducing the intensity of oppositional behaviour and aggressiveness and allowing a diminution of neuroleptic treatment.

DETAILED DESCRIPTION:
A technique of receptive music therapy to induce relaxation has been developed in the university hospital of Montpellier: the "U" sequence. The musical sequence lasts 20 minutes and is made up of several phases that progressively induce a relaxed state in the patient. This effect is obtained by modulating the rhythm of the music, the orchestral formation, frequencies and volume. The phase of maximum relaxation is followed by a stimulating phase. These musical sequences have been specially designed by the music publishers Music Care©.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either sex aged 65 years and over, living in an institution for the dependent elderly for at least 3 months
* Subjects with Alzheimer-type dementia (DSM-IV and National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria)or related symptoms
* If treated, Treated for at least 6 months with a stable dose of cholinesterase inhibitor or memantine
* Mini-Mental State Examination (MMSE) score between 5 and 20
* Patients with disruptive behaviour (at least one disruptive item on the NPI: oppositional behaviour/aggressiveness/agitation, aberrant motor behaviour, with a severity score grater than or equal to 4) and treated with at least one neuroleptic whose dose which could not be decreased because of persistence of the behavioural problems for at least 15 days.

Exclusion Criteria:

* Decompensated physical disease
* Inability to give informed consent
* Lack of health insurance coverage
* Non-corrected hearing impairment
* treatment ongoing with two or more neuroleptics

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Neuroleptic reduction dose | during 2 months
  Benefit obtained in terms of the reduction in neuroleptic dose

SECONDARY OUTCOMES:
Durability of treatment effect | 1, 2 and 3 months
  Score on the Cohen-Mansfield scale, Overall NPI score, Quality of life in Alzheimer's disease scale (QOL-AD)

OTHER OUTCOMES:
Music therapy session's effects | 4 weeks after completion of music therapy sessions
  Proportions of patients in the two groups who discontinued neuroleptics, Scores on the Cohen-Mansfield scale, Dose of neuroleptics

CONTACTS AND LOCATIONS:
Overall Officials: Christophe ARBUS, MD, Principal Investigator — University Hospital, Toulouse
Locations (7):
- France (7):
  - University Hospital Toulouse, Toulouse, Midi-Pyrenees
  - EHPAD La Villegiale, Castres, Tarn
  - Residence Christian Bressole, Castres, Tarn
  - EHPAD L'Oustal d'en Thibaud, Labruguière, Tarn
  - EHPAD Les Quietudes, Lautrec, Tarn
  - EHPAD KORIAN Grand Maison, L'Union
  - Centre Hospitalier Gérard Marchant, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aalten P, de Vugt ME, Jaspers N, Jolles J, Verhey FR. The course of neuropsychiatric symptoms in dementia. Part I: findings from the two-year longitudinal Maasbed study. Int J Geriatr Psychiatry. 2005 Jun;20(6):523-30. doi: 10.1002/gps.1316. PMID 15920712
- [Background] Aldridge D. Music and Alzheimer's disease--assessment and therapy: discussion paper. J R Soc Med. 1993 Feb;86(2):93-5. No abstract available. PMID 8433315
- [Background] Benoit M, Robert PH, Staccini P, Brocker P, Guerin O, Lechowski L, Vellas B; REAL.FR Group. One-year longitudinal evaluation of neuropsychiatric symptoms in Alzheimer's disease. The REAL.FR Study. J Nutr Health Aging. 2005;9(2):95-9. PMID 15791352
- [Background] Cohen-Mansfield J, Marx MS, Rosenthal AS. A description of agitation in a nursing home. J Gerontol. 1989 May;44(3):M77-84. doi: 10.1093/geronj/44.3.m77. PMID 2715584
- [Derived] van der Steen JT, van der Wouden JC, Methley AM, Smaling HJA, Vink AC, Bruinsma MS. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2025 Mar 7;3(3):CD003477. doi: 10.1002/14651858.CD003477.pub5. PMID 40049590